CLINICAL TRIAL: NCT01880255
Title: Repetitive Transcranial Magnetic Stimulation (rTMS) for the Treatment of Working Memory Deficits in Schizophrenia and Effects on Brain Structure
Brief Title: rTMS for Working Memory Deficits in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Aristotle Voineskos, Director, Slaight Family Centre for Youth in Transition; Head, Kimel Family Imaging-Genetics Laboratory, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 057/2013
Record Dates: First submitted 2013-06-14; First posted 2013-06-18 (Estimated); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Repetitive Transcranial Magnetic Stimulation; Schizophrenia; Cognition; Working Memory
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active rTMS (Active Comparator): Active treatment will be delivered at an intensity that is 90% of the resting motor threshold (RMT). Stimulation will be delivered at 20 Hz with 25 stimulation trains of 30 stimuli each (i.e., 750 stimuli) and an intertrain interval of 30 sec. Treatment will be applied in sequential order bilaterally to the left and right dorsolateral prefrontal cortex (DLPFC). The order of bilateral stimulation (i.e. right then left or left then right) will be held constant for all 20 treatments.
  Intervention: Device: Repetitive Transcranial Magnetic Stimulation
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- Sham rTMS (Sham Comparator): Sham stimulation will be delivered using the same stimulation parameters and at the site of active treatment, but with only the side-edge resting on the scalp. The coil will be angled 45 degrees away from the skull in a single-wing tilt position. This method produces sound and some somatic sensation (e.g., contraction of scalp muscles) similar to those of active stimulation, but with minimal direct brain effects.
  Intervention: Device: Repetitive Transcranial Magnetic Stimulation
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — rTMS is a non-invasive procedure involving the use of magnetic fields to stimulate nerve cells.
  Other Names: MagPro X100 Series (Medtronic A/S, Copenhagen, Denmark)

SUMMARY:
In this study, the investigators will be examining the effects of repetitive transcranial magnetic stimulation (rTMS) on memory deficits in individuals with schizophrenia and schizoaffective disorder. Half of the study participants will be chosen by chance to receive active rTMS stimulation while half will be chosen by chance to receive sham rTMS. Sham rTMS will feel the same as active rTMS only there will be no direct brain stimulation. This is necessary to ensure that active rTMS is efficacious in the enhancement of memory in individuals with schizophrenia. Based on results from a recently published pilot study, the investigators propose that active rTMS treatment will result in a significant improvement in working memory performance compared to sham rTMS treatment.

DETAILED DESCRIPTION:
This study is a randomized, double blind, sham controlled study to evaluate the efficacy of repetitive transcranial magnetic stimulation as a treatment for working memory deficits in individuals with schizophrenia or schizoaffective disorder between 18 and 59 years of age. The study duration is approximately 3 months, with the rTMS sessions lasting for 4 weeks, 5 times a week, for about 1 hour each. Several scales will be used to assess symptom severity as part of the clinical assessment. Cognition will be assessed using a validated battery and the N-back task.

This study also involves a type of brain imaging known as magnetic resonance imaging (MRI) at the beginning and at the end of the 4 weeks of daily rTMS to better understand the effects of rTMS on brain structure and function. Investigators will measure the size and connections of different parts of the brain to assess brain structure and blood flow while you are completing some basic tasks to assess brain function. We will also collect two blood samples (before and after rTMS treatment) to see if certain proteins change in response to treatment. Finally, an analysis of genetic material will be conducted to see if genes play a role in differences in how people respond to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 59 years of age
* Current diagnosis of Schizophrenia or Schizoaffective Disorder
* Able to provide written informed consent
* Fluency in the English Language

Exclusion Criteria:

* Have a history of substance abuse or dependence in the last 6 months
* Have a concomitant major and unstable medical or neurologic illness
* Have a history of seizures or have a first degree relative with a history of a seizure disorder
* Current pregnancy or a plan to become pregnant during the duration of the study
* Clinical instability: determined by treating physician
* Have received electroconvulsive therapy (ECT) within the last year
* Have a history of repetitive transcranial magnetic stimulation (rTMS)
* Are taking a benzodiazepine at a dose greater than Lorazepam 2mg or equivalent
* Are taking any non-benzodiazepine anticonvulsant
* Have a cardiac pacemaker, cochlear implant, implanted electronic device or non-electric metallic implant

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2013-06; Primary Completion 2019-01-07 (Actual); Study Completion 2019-01-07 (Actual)

PRIMARY OUTCOMES:
Performance on the N-back working memory task | 4 weeks
  The primary outcome measure will be the performance on the N-back working memory task. Specifically, we will evaluate if rTMS results in a change in percent of correct responses in the N-back task.
  Note: the N-back is a continuous performance task that is commonly used to measure attention and working memory.

SECONDARY OUTCOMES:
Brain Imaging Changes | 4 weeks
  For brain imaging we will test for group differences using: (1) cortical thickness (2) volumetric measures, (3) diffusion based measures. Statistical tests measuring these differences will be conducted at baseline and following the final rTMS treatment session. We will control for possible effects of neuroleptic medication on MRI measures by regressing mean dosage levels multiplied by number of years on medication, for each of five classes of medication (typical neuroleptics, atypical neuroleptics, antiparkinsonian anticholinergics, lithium, benzodiazepines)

CONTACTS AND LOCATIONS:
Overall Officials: Aristotle Voineskos, MD, PHD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Voineskos AN, Blumberger DM, Schifani C, Hawco C, Dickie EW, Rajji TK, Mulsant BH, Foussias G, Wang W, Daskalakis ZJ. Effects of Repetitive Transcranial Magnetic Stimulation on Working Memory Performance and Brain Structure in People With Schizophrenia Spectrum Disorders: A Double-Blind, Randomized, Sham-Controlled Trial. Biol Psychiatry Cogn Neurosci Neuroimaging. 2021 Apr;6(4):449-458. doi: 10.1016/j.bpsc.2020.11.011. Epub 2020 Nov 28. PMID 33551284
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching hospital. It is fully affiliated with the University of Toronto, and is a PAHO/WHO Collaborating Centre — http://www.camh.net/research